CLINICAL TRIAL: NCT04004195
Title: Investigation of Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of a Single Oral Dose of BAY2327949 Given as Immediate Release Tablet in Male and Female Participants in a Multi-center, Non-randomized, Non-controlled, Non-blinded Study With Group Stratification in Participants With Renal Impairment and Healthy Participants Matched for Age, Gender, and Weight
Brief Title: Study to Investigate Safety, Absorption, Elimination, and Drug Effect of BAY2327949 in Participants With Different Renal Function Status
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19224; 2019-000630-19 (EudraCT Number)
Record Dates: First submitted 2019-06-28; First posted 2019-07-01 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy participants (Experimental)
  Interventions: Drug: BAY2327949
- Participants with mild renal impairment (Experimental)
  Interventions: Drug: BAY2327949
- Participants with moderate renal impairment (Experimental)
  Interventions: Drug: BAY2327949
- Participants with severe renal impairment (Experimental)
  Interventions: Drug: BAY2327949

INTERVENTIONS:
Drug: BAY2327949 — A single oral dose of 30 mg BAY2327949 given as one 30 mg IR tablet (dose might be reduced to 15 mg for group 4 according to safety assessment team decision)

SUMMARY:
BAY2327949 is currently under clinical development for chronic kidney disease. The goal of this study is to learn more about how the body absorbs, distributes and excretes the study drug when taken once per mouth as 30mg tablet. An additional important goal of this study is to gain more information on how well the study drug is tolerated and its effect on the human body functions. The study will enroll healthy participants or patients with mild, moderate or severe reduced kidney functions matched for age, weight and gender. The results of this study will help researchers to select the best dosing of the study drug for future studies in patients.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥18 years of age
* The study enrolls healthy participants and participants at different stages of renal impairment (mild to severe renal impairment).
* Race: White
* BMI (body mass index): above or equal 18.5 and below or equal 35 kg/m*2 at the first screening visit.
* Male or female.
* Participants with renal impairment must have an eGFR (estimated glomerular filtration rate) <90 mL/min/1.73 m*2 determined from serum creatinine 21-3 days prior to dosing using the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) equation (eGFR has to be repeated if screening period >10 days before dosing).

Stable renal function, e.g. a serum creatinine value determined at least 3 months before the pre-study visit should not vary by more than 25% from the serum creatinine value determined at the pre-study visit confirmed by nephrologist or general practitioner the patient is under care.

Exclusion Criteria:

* Clinically relevant findings in the physical examination affecting the objectives of the study.
* Systemic use of the following co-medications from 2 weeks before administration until end of follow-up:

  * Moderate and strong inhibitors of CYP3A;
  * Moderate and strong CYP3A inducers;
  * Moderate and strong inhibitors of P-gp transport;
  * UDP-glucuronosyltransferase (UGT) inhibitors probenecid and valproic acid.
* Regular daily consumption of more than 10 cigarettes.
* Acute renal failure.
* Active nephritis.
* Impairment of any other major organ system other than the kidney.
* Change in chronic medications for renal disease (or its consequences) less than 4 weeks prior to dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Cmax of BAY2327949 | From pre-dose until follow-up (10-12 days after dosing).
  Cmax: Maximum observed drug concentration in measured matrix after single dose administration
AUC of BAY2327949 | From pre-dose until follow-up (10-12 days after dosing).
  AUC:Area under the concentration vs. time curve from zero to infinity after single (first) dose.
  AUC(0-tlast) will be used as primary variables if mean AUC(tlast-∞) >20% of AUC
Cmax,u of BAY2327949 | From pre-dose until follow-up (10-12 days after dosing).
  Cmax,u: Cmax based on the unbound plasma concentrations of the study drug
AUCu of BAY2327949 | From pre-dose until follow-up (10-12 days after dosing).
  AUC(0-tlast)u will be used as primary variables if mean AUC(tlast-∞) >20% of AUC

SECONDARY OUTCOMES:
Frequency and nature of treatment-emergent adverse events | Approximate 14 days (from starting treatment to end of follow-up)
Urinary volume | From Day -1 until Day 4 (72h after dosing)
Fluid balance | From Day -1 until Day 4 (72h after dosing)

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - APEX GmbH, München, Bavaria
  - CRS Clinical-Research-Services Kiel GmbH, Kiel, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.